CLINICAL TRIAL: NCT03782688
Title: Prospective Evaluation of a Virtual Non-invasive Percutaneous Intervention Planner in Patients With Coronary Artery Disease.
Brief Title: Precise Percutaneous Coronary Intervention Plan (P3) Study
Acronym: P3
Status: Completed | Type: Observational
Sponsor: Onze Lieve Vrouw Hospital (Other)
Responsible Party: Principal Investigator, Jeroen Sonck, Co-Director Cardiovascular Center OLV-Aalst, Onze Lieve Vrouw Hospital
Other Study IDs: CVBA-CRI_0001
Record Dates: First submitted 2018-12-12; First posted 2018-12-20 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Stable Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single-arm cohort: Patients with significant coronary stenosis by invasive fractional flow reserve (FFR≤0.80)
  Interventions: Diagnostic Test: FFRCT planner

INTERVENTIONS:
Diagnostic Test: FFRCT planner — Non-invasive post-PCI fractional flow reserve prediction
  Other Names: HeartFlow Planner

SUMMARY:
The PRECISE PERCUTANEOUS CORONARY INTERVENTION (PCI) PLAN STUDY is an investigator-initiated, international and multicenter study of patients with an indication for PCI aiming at assessing the agreement and accuracy of the HeartFlow Planner with invasive fractional flow reserve (FFR) as a reference.

DETAILED DESCRIPTION:
Multicenter study, including 120 patients at 5 centers in Europe and Asia. After identifying the presence of significant coronary stenosis by means of coronary angiography and invasive fractional flow reserve (FFR≤0.80) the patients will undergo the following procedures: Invasive FFR with intravenous adenosine (i.e. pre- and post-PCI). Optical coherence tomography-guided PCI (i.e. pre- and post-procedural imaging). PCI with newer generation drug-eluting stent.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease in a major epicardial vessel with an invasive fractional flow reserve (FFR) ≤0.80
* An indication to Percutaneous coronary intervention

Exclusion Criteria:

- Angiographic exclusion criteria

1. Severely calcified lesion/vessel
2. Bifurcation lesions.
3. Ostial lesions.
4. Left main disease.
5. Severe vessel tortuosity.

Clinical exclusion criteria

1. Chronic obstructive pulmonary disease
2. Contraindication to adenosine
3. NYHA class III or IV, or last known left ventricular ejection fraction <30%
4. Uncontrolled or recurrent ventricular tachycardia
5. Atrial fibrillation, flutter or arrhythmia
6. History of recent stroke (≤90 days)
7. History of acute coronary syndrome (≤90 days)
8. Prior myocardial infarction
9. History of ischemic stroke (>90 days) with modified RANKIN score ≥ 2
10. History of any hemorrhagic stroke
11. Previous revascularization (PCI or Coronary artery bypass grafting)
12. Active liver disease or hepatic dysfunction, defined as AST or ALT > 3 times the ULN
13. Severe renal dysfunction, defined as an eGFR <30 mL/min/1.73 m2
14. Body mass index>35 kg/m2
15. Nitrate intolerance
16. Contra-indication to heart rate lowering drugs

    Imaging-related
17. Insufficient coronary CT Angiography image quality.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Stable Coronary Artery Disease with Positive Fractional Flow Reserve and indication for percutaneous myocardial revascularization.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
Agreement on post-PCI fractional flow reserve between virtual treatment based on FFRct planner and measured invasive post-PCI fractional flow reserve. | The primary endpoint will be assessed immediately after the procedure (PCI).
  The agreement will be assessed by Bland Altman method

CONTACTS AND LOCATIONS:
Overall Officials: Bernard De Bruyne, MD, PhD, Study Chair — OLV-Aalst
Locations (1):
- OLV-Aalst, Aalst, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Undecided plan for data sharing

REFERENCES:
- [Derived] Seki R, Collison D, Ikeda K, Sonck J, Munhoz D, Bertolone DT, Ko B, Maeng M, Otake H, Koo BK, Storozhenko T, Bouisset F, Belmonte M, Leone A, Shumkova M, Ford TJ, Mahendiran T, Berry C, De Bruyne B, Oldroyd K, Sakai K, Mizukami T, Collet C. Validation of virtual fractional flow reserve pullback curves. Catheter Cardiovasc Interv. 2024 Nov;104(6):1178-1188. doi: 10.1002/ccd.31222. Epub 2024 Sep 29. PMID 39342486
- [Derived] Yang S, Hwang D, Sakai K, Mizukami T, Leipsic J, Belmonte M, Sonck J, Norgaard BL, Otake H, Ko B, Maeng M, Moller Jensen J, Buytaert D, Munhoz D, Andreini D, Ohashi H, Shinke T, Taylor CA, Barbato E, De Bruyne B, Collet C, Koo BK. Predictors for Vulnerable Plaque in Functionally Significant Lesions. JACC Cardiovasc Imaging. 2025 Feb;18(2):195-206. doi: 10.1016/j.jcmg.2024.07.021. Epub 2024 Sep 11. PMID 39269415
- [Derived] Candreva A, Gallo D, Munhoz D, Rizzini ML, Mizukami T, Seki R, Sakai K, Sonck J, Mazzi V, Ko B, Norgaard BL, Jensen JM, Maeng M, Otake H, Koo BK, Shinke T, Aben JP, Andreini D, Gallinoro E, Stahli BE, Templin C, Chiastra C, De Bruyne B, Morbiducci U, Collet C. Influence of intracoronary hemodynamic forces on atherosclerotic plaque phenotypes. Int J Cardiol. 2024 Mar 15;399:131668. doi: 10.1016/j.ijcard.2023.131668. Epub 2023 Dec 22. PMID 38141723
- [Derived] Sakai K, Mizukami T, Leipsic J, Belmonte M, Sonck J, Norgaard BL, Otake H, Ko B, Koo BK, Maeng M, Jensen JM, Buytaert D, Munhoz D, Andreini D, Ohashi H, Shinke T, Taylor CA, Barbato E, Johnson NP, De Bruyne B, Collet C. Coronary Atherosclerosis Phenotypes in Focal and Diffuse Disease. JACC Cardiovasc Imaging. 2023 Nov;16(11):1452-1464. doi: 10.1016/j.jcmg.2023.05.018. Epub 2023 Jul 19. PMID 37480908
- [Derived] Mizukami T, Sonck J, Sakai K, Ko B, Maeng M, Otake H, Koo BK, Nagumo S, Norgaard BL, Leipsic J, Shinke T, Munhoz D, Mileva N, Belmonte M, Ohashi H, Barbato E, Johnson NP, De Bruyne B, Collet C. Procedural Outcomes After Percutaneous Coronary Interventions in Focal and Diffuse Coronary Artery Disease. J Am Heart Assoc. 2022 Dec 6;11(23):e026960. doi: 10.1161/JAHA.122.026960. Epub 2022 Nov 29. PMID 36444858
- [Derived] Sonck J, Nagumo S, Norgaard BL, Otake H, Ko B, Zhang J, Mizukami T, Maeng M, Andreini D, Takahashi Y, Jensen JM, Ihdayhid A, Heggermont W, Barbato E, Mileva N, Munhoz D, Bartunek J, Updegrove A, Collinsworth A, Penicka M, Van Hoe L, Leipsic J, Koo BK, De Bruyne B, Collet C. Clinical Validation of a Virtual Planner for Coronary Interventions Based on Coronary CT Angiography. JACC Cardiovasc Imaging. 2022 Jul;15(7):1242-1255. doi: 10.1016/j.jcmg.2022.02.003. Epub 2022 Apr 13. PMID 35798401